CLINICAL TRIAL: NCT06092931
Title: A Phase 1, Single-Center, Open-Label, Fixed-Sequence Study to Evaluate the Effect of DC-806 on the Single Dose Pharmacokinetics of CYP450 Enzyme and Transporter Substrates in Healthy Participants
Brief Title: A Drug-Drug Interaction Study Evaluating the Perpetrator Potential of DC-806 on Cocktails of CYP450 Enzyme and Transporter Substrates in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCE806104
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy Participants
Keywords: DC-806; Drug-drug interaction; Midazolam; Repaglinide; Digoxin; Rosuvastatin
MeSH Terms: interventions — Midazolam; repaglinide; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: DC-806 + Midazolam (CYP3A4 substrate) + Repaglinide (CYP2C8 substrate) (Experimental): Participants will receive a single oral dose of the 2-probe substrate cocktail (midazolam and repaglinide) on Day 1. From Day 4 through Day 8, participants will receive twice-daily (BID) oral doses of DC-806 and a single oral dose of the 2-probe substrate cocktail on Day 7. DC-806 BID dosing will continue until the end of Day 8.
  Interventions: Drug: DC-806; Drug: Midazolam; Drug: Repaglinide
- Cohort 2: DC-806 + Digoxin (P-gp substrate) + Rosuvastatin (BCRP/OATP1B1 substrate) (Experimental): Participants will receive a single oral dose of the 2-probe substrate cocktail (digoxin and rosuvastatin) on Day 1. From Day 5 through Day 9, participants will receive twice daily oral doses of DC-806 and a single oral dose of the 2-probe substrate cocktail on Day 8. DC-806 BID dosing will continue until the end of Day 9.
  Interventions: Drug: DC-806; Drug: Digoxin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: DC-806 — Oral tablets
Drug: Midazolam — Oral syrup
  Arms: Cohort 1: DC-806 + Midazolam (CYP3A4 substrate) + Repaglinide (CYP2C8 substrate)
Drug: Repaglinide — Oral tablets
  Arms: Cohort 1: DC-806 + Midazolam (CYP3A4 substrate) + Repaglinide (CYP2C8 substrate)
Drug: Digoxin — Oral tablets
  Arms: Cohort 2: DC-806 + Digoxin (P-gp substrate) + Rosuvastatin (BCRP/OATP1B1 substrate)
Drug: Rosuvastatin — Oral tablets
  Arms: Cohort 2: DC-806 + Digoxin (P-gp substrate) + Rosuvastatin (BCRP/OATP1B1 substrate)

SUMMARY:
The main objective of this study is to assess the effect of DC-806 on the pharmacokinetics (PK) of cytochrome 3A4 (CYP3A4) substrate, midazolam and its active metabolite, 1-hydroxymidazolam, cytochrome 2C8 (CYP2C8) substrate repaglinide, P-glycoprotein (P-gp) transporter substrate digoxin, and breast cancer resistant protein (BCRP)/ organic anion transporter protein-1B1 (OATP1B1) transporter substrate rosuvastatin in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male or female; females must be of nonchildbearing potential, or postmenopausal.
2. Age: 18 to 55 years, inclusive, at screening.
3. Body mass index: 18.0 to 32.0 kg/m^2, inclusive, at screening.
4. Weight: ≥50 kg at screening.
5. Status: healthy participants.
6. At screening, females must be of nonchildbearing potential (defined as at least 12 consecutive months with no menses prior to screening, a serum follicle-stimulating hormone test to confirm postmenopausal status, or being surgically sterilized); nonpregnancy will be confirmed for all females by a serum pregnancy test conducted at screening, and by a urine pregnancy test at admission and at follow-up.
7. Male participants, if not permanently surgically sterilized, must inform all sexual partners of their participation in a research study and agree to use a highly effective method of contraception and not donate sperm from admission to the clinical site until 30 days after the last study drug administration.
8. All prescribed medication must have been stopped at least 14 days prior to admission to the clinical site.
9. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (e.g., St. John's wort) must have been stopped at least 7 days (or 5 half-lives for certain medications, whichever is longer) prior to admission to the clinical site. Occasional use of acetaminophen/paracetamol (e.g., up to 2 grams per day) is permitted during this period and throughout the study.
10. Ability and willingness to abstain from alcohol-, caffeine-, and methylxanthine- containing beverages or food (e.g., coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to admission to the clinical site and during confinement at the clinical site.
11. Willingness to abstain from any strenuous physical exercise from 96 hours (4 days) prior to admission and during confinement at the clinical site.
12. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory assessments, 12-lead electrocardiograms, and vital signs, as judged by the Investigator.
13. Willing and able to sign the informed consent form.

Exclusion Criteria:

1. Employee of Contract Research Organization or the Sponsor.
2. History of relevant drug and/or food allergies, in the opinion of the Investigator.
3. Females who are currently breastfeeding.
4. Smoking more than 5 cigarettes, 1 cigar, or 1 pipe daily within 3 months prior to screening.
5. Unwilling or unable to abstain from tobacco products within the 48 hours (2 days) prior to admission and during confinement in the clinical site.
6. History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within 1 year prior to screening.
7. Positive drug and/or alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening or admission to the clinical site.
8. History within the previous 12 months of alcohol consumption exceeding 2 standard drinks per day on average. Alcohol consumption will be prohibited 48 hours prior to admission to the clinical site and during confinement at the clinical site.
9. Positive screen for hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency virus 1 and 2 antibodies.
10. Consumption of any nutrients known to modulate CYP450 enzymes activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to the first administration of study drug and during the study (including washout period/clinic furlough until after discharge in the last study period).
11. Participation in a drug study within 30 days prior to study drug administration in the current study. Participation in 4 or more other drug studies in the 12 months prior to study drug administration in the current study.
12. History of donation of more than 450 mL of blood within 60 days prior to dosing in the clinical site or planned donation before 30 days has elapsed since intake of study drug.
13. Plasma or platelet donation within 7 days of dosing and through follow-up.
14. Significant and/or acute illness within 5 days prior to study drug administration that may impact safety assessments, in the opinion of the Investigator.
15. Unsuitable veins for infusion or blood sampling as determined by the Investigator or study staff.
16. Any other condition or prior therapy that, in the Investigator's opinion, would confound or interfere with the evaluation of safety, tolerability, or PK of the study drug, interfere with study compliance, or preclude informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Maximum Observed Plasma Concentration (Cmax) of Midazolam | Day 1 and Day 7
Cohort 1: Cmax of 1-hydroxymidazolam | Day 1 and Day 7
Cohort 1: Cmax of Repaglinide | Day 1 and Day 7
Cohort 2: Cmax of Digoxin | Day 1 and Day 8
Cohort 2: Cmax of Rosuvastatin | Day 1 and Day 8
Cohort 1: Area Under the Plasma Concentration-time Curve (AUC) up to Time t, Where t is the Last Point with Concentrations Above the Lower Limit of Quantification (AUC0-t) of Midazolam | Days 1-3 and Days 7-9
Cohort 1: AUC0-t of 1-hydroxymidazolam | Days 1-3 and Days 7-9
Cohort 1: AUC0-t of Repaglinide | Days 1-3 and Days 7-9
Cohort 2: AUC0-t of Digoxin | Days 1-5 and Days 8-12
Cohort 2: AUC0-t of Rosuvastatin | Days 1-5 and Days 8-12
Cohort 1: AUC from Time 0 to Infinity (AUC0-inf) of Midazolam | Days 1-3 and Days 7-9
Cohort 1: AUC0-inf of 1-hydroxymidazolam | Days 1-3 and Days 7-9
Cohort 1: AUC0-inf of Repaglinide | Days 1-3 and Days 7-9
Cohort 2: AUC0-inf of Digoxin | Days 1-5 and Days 8-12
Cohort 2: AUC0-inf of Rosuvastatin | Days 1-5 and Days 8-12

SECONDARY OUTCOMES:
Cohorts 1 and 2: Number of Participant who Experience an Adverse Event | Up to a maximum 22 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Phase 1 Clinic, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No